CLINICAL TRIAL: NCT00000901
Title: A Multicenter, Open-Labeled, 96-Week Study to Investigate the Safety, Pharmacokinetics, and Efficacy of Indinavir in Combination With Stavudine and Lamivudine in Pediatric Patients With HIV-1 Infection
Brief Title: Safety and Effectiveness of Giving Indinavir Plus Stavudine Plus Lamivudine to HIV-Infected Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 395; 11351 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Dose-Response Relationship, Drug; Drug Therapy, Combination; Stavudine; HIV Protease Inhibitors; Lamivudine; Indinavir; RNA, Viral; Reverse Transcriptase Inhibitors; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Lamivudine; Stavudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Lamivudine
Drug: Stavudine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give an anti-HIV drug combination of indinavir (IDV) plus stavudine (d4T) plus lamivudine (3TC) to HIV-infected children. IDV will be given either as a powder mixed into applesauce or as capsules given on an empty stomach.

DETAILED DESCRIPTION:
In this multicenter, open-label study patients receive a combined drug regimen of indinavir, stavudine, and lamivudine over 48 weeks. Patients are evaluated at Weeks 0, 2, 4, every 4 weeks until Week 24, and every 8 weeks thereafter until study completion. [AS PER AMENDMENT 4/27/99: The study has been extended for an additional 48 weeks for a total of 96 weeks.]

ELIGIBILITY:
Inclusion Criteria

Your child may be eligible for this study if he/she:

* Is 3 - 15 years old and has consent of a parent or legal guardian who is able to return with the child for follow-up visits.
* Is HIV-positive.
* Is generally healthy.
* Is able to swallow medication in capsule form.
* Has never taken d4T or has never taken 3TC.
* Agrees to use barrier methods of birth control (such as condoms) during the study. The pill is not allowed during the study.

Exclusion Criteria

Your child will not be eligible for this study if he/she:

* Has a serious infection at the time of study entry.
* Has a history of severe diarrhea.
* Is unable to take any of the medications in this study for any reason.
* Has a history of certain serious illnesses.
* Has taken any protease inhibitors (PIs).
* Has taken any non-nucleoside reverse transcriptase inhibitors (NNRTIs), such as efavirenz (EFV), within 2 weeks prior to study entry.
* Has taken certain medications.
* Is pregnant or breast-feeding.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24
Dates: Study Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Sleasman, Study Chair; Ross McKinney, Study Chair
Locations (19):
- United States (18):
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Yale Univ Med School, New Haven, Connecticut
  - Univ of Florida Gainesville, Gainesville, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Children's Hosp of Boston, Boston, Massachusetts
  - North Shore Univ Hosp, Great Neck, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- San Juan City Hosp, San Juan, Puerto Rico